CLINICAL TRIAL: NCT01707667
Title: An Open-label, Randomized, Crossover, Reader-blinded Study to Investigate the Effect of Prucalopride and Polyethylene Glycol 3350 on Colon Motility With Intramural Manometry in Subjects With Chronic Constipation
Brief Title: Study to Investigate Prucalopride vs. Polyethylene Glycol 3350 on Colon Activity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SPD555-403; 2012-002495-13 (EudraCT Number)
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Chronic Constipation
MeSH Terms: interventions — prucalopride; polyethylene glycol 3350

ARMS (2):
- Prucalopride (Experimental)
  Interventions: Drug: prucalopride
- PEG 3350 (Active Comparator)
  Interventions: Drug: PEG 3350

INTERVENTIONS:
Drug: prucalopride — One 2 mg tablet orally administered on Day 1
  Other Names: Resolor (Marketed name in Europe)
  Arms: Prucalopride
Drug: PEG 3350 — 13.8g polyethylene glycol (PEG) 3350 with sodium bicarbonate, sodium chloride, and potassium chloride as a solution in water. Administered twice orally on Day 1(once in the morning and once prior to lunch).
  Other Names: Movicol
  Arms: PEG 3350

SUMMARY:
To evaluate the different effects of prucalopride and PEG 3350 + electrolytes on colon motor activity in subjects that are chronically constipated.

ELIGIBILITY:
Inclusion Criteria:

* Chronic constipation
* Male or female ages 18-75 years
* Non-pregnant, non-lactating female

Exclusion Criteria:

* Drug-induced constipation
* Subjects suffering from secondary causes of chronic constipation, such as:
* Endocrine disorders, e.g. hypopituitarism, hypothyroidism, hypercalcemia, pseudohypoparathyroidism, pheochromocytoma or glucagon-producing tumors, unless these are controlled by appropriate medical therapy.
* Metabolic disorders, e.g. porphyria, uremia, hypokalemia or amyloid neuropathy, unless these are controlled by appropriate medical therapy
* Neurological disorders, e.g. Parkinson's disease, cerebral tumors, cerebrovascular accidents, multiple sclerosis, meningocele, aganglionosis, hypoganglionosis, hyperganglionosis, autonomic neuropathy or neuropathy due to chemotherapy, spinal cord injury, Chaga's disease, or major depression
* Surgery.
* Subjects with insulin-dependent diabetes mellitus
* Rectal evacuation disorder/outlet obstruction
* Subjects with intestinal perforation or obstruction
* Severe renal impairment
* Subjects with a history of alcohol or drug abuse
* Subjects with lactose intolerance
* Subjects with clinically significant cardiac, vascular, liver, pulmonary, endocrine, neurological or psychiatric disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-02-27 (Actual); Primary Completion 2013-11-27 (Actual); Study Completion 2013-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma, United States
- UNIVERSITY OF LEUVEN, UNVERSITY HOSPITAL, Gasthuisberg, Leuven, Belgium
- Barts Health NHS Trust, Whitechapel, London, United Kingdom

REFERENCES:
- [Derived] Miner PB Jr, Camilleri M, Burton D, Achenbach H, Wan H, Dragone J, Mellgard B. Prucalopride induces high-amplitude propagating contractions in the colon of patients with chronic constipation: a randomized study. Neurogastroenterol Motil. 2016 Sep;28(9):1341-8. doi: 10.1111/nmo.12832. Epub 2016 Jun 7. PMID 27270968

RESULTS

PARTICIPANT FLOW:
Groups:
- PRU-PEG: A single dose of prucalopride 2mg in the first period followed by 2 doses of polyethylene glycol (PEG) 3350 (13.8g) plus electrolytes in the second period.
- PEG-PRU: Two doses of PEG 3350 (13.8g) plus electrolytes in the first period followed by a single dose of prucalopride 2mg in the second period.
Period: Period 1
Arm/Group | PRU-PEG | PEG-PRU
Started | 7 | 6
Completed | 6 | 6
Not Completed | 1 | 0
Not completed — expulsion of colonic sensor catheter | 1 | 0
Period: Period 2
Arm/Group | PRU-PEG | PEG-PRU
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set consisted of all randomized subjects who had taken at least 1 dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | PRU-PEG | PEG-PRU | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.3 (11.04) | 35.2 (13.18) | 37.9 (11.85)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 | 7 | 6 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: The Number of High-Amplitude Propagating Contractions (HAPC)
Description: Manometry recordings were read by an experienced gastroenterologist who was blinded to the treatment each subject received. The tracings were analyzed using computer-based validated software. HAPC and manometry data were available for every sensor as well as average values for each HAPC and manometry time point. The primary outcome analysis of HAPC data used the following threshold: Mean amplitude ≥100mmHg and extension ≥20cm (9 sensors).
Time Frame: over 12 hours post-dose
Population: The Pharmacodynamic Analysis Set consisted of all randomized subjects who had taken at least 1 dose of investigational product and who had 1 evaluable manometry assessment (minimum of 4 hours of manometry recordings from the intake of investigational product) for each treatment period.
Measure: Least Squares Mean (Standard Error); unit: Number of HAPC with amplitude ≥100mmHg
Groups:
- Prucalopride: A single dose of 2mg prucalopride, administered orally as tablets with 125mL of water on Day 1.
- PEG 3350: 13.8g polyethylene glycol (PEG) 3350 with sodium bicarbonate, sodium chloride, and potassium chloride as a solution in water. Administered twice orally on Day 1 (once in the morning and once prior to lunch).
Arm/Group | Prucalopride | PEG 3350
Number analyzed (Participants) | 12 | 12
Number of HAPC with amplitude ≥100mmHg | 8.7 (2.06) | 2.9 (2.06)
Statistical Analysis 1: Comparison: Prucalopride vs PEG 3350; Test type: Superiority or Other; p = 0.012, Linear Mixed-Effect Models Analysis; Mean Difference (Final Values) = 5.8, 95% CI 2-sided [1.6 to 9.9]

2. Secondary Outcome: Area Under the Concentration Curve (AUC) of All HAPCs
Description: The AUC of all HAPCs during the first 12 hours after treatment was calculated as the sum of the AUC at all sensors of each HAPC at the ≥100mmHg and ≥20cm threshold.
Time Frame: over 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg.sec
Arm/Group | Prucalopride | PEG 3350
Number analyzed (Participants) | 9 | 6
mmHg.sec | 110204.1 (28279.91) | 41152.7 (34432.61)
Statistical Analysis 1: Comparison: Prucalopride vs PEG 3350; Test type: Superiority or Other; p = 0.079, Linear Mixed-Effect Models Analysis; Mean Difference (Final Values) = 69051.4, 95% CI 2-sided [-12004.5 to 150107.3]

3. Secondary Outcome: The Mean Amplitude of HAPC
Description: The mean amplitude of all HAPCs was calculated as the sum of the mean amplitude for each HAPC divided by the number of HAPCs.
Time Frame: over 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Prucalopride | PEG 3350
Number analyzed (Participants) | 9 | 6
mmHg | 199.0 (15.15) | 189.8 (19.56)
Statistical Analysis 1: Comparison: Prucalopride vs PEG 3350; Test type: Superiority or Other; p = 0.717, Linear Mixed-Effect Models Analysis; Mean Difference (Final Values) = 9.2, 95% CI 2-sided [-45.3 to 63.7]

4. Secondary Outcome: Time to First HAPC
Description: The median (95% CI) time to first HAPC after administration of investigational product with amplitude ≥100mmHg and extension ≥20cm.
Time Frame: over 12 hours post-dose
Population: The Pharmacodynamic Analysis Set included all subjects in the Safety Analysis Set who had 1 evaluable manometry assessment (minimum of 4 hours of manometry recordings from the intake of investigational product) for each treatment period.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Prucalopride | PEG 3350
Number analyzed (Participants) | 9 | 6
hours | 4.5 [1.5 to 9.3] | NA [2.8 to NA] — The median time to first HAPC after administration of investigational product with amplitude ≥100mmHg and extension ≥20cm in the PEG 3350 group could not be calculated as only 6 subjects had HAPCs that met this threshold.
Statistical Analysis 1: Comparison: Prucalopride vs PEG 3350; Test type: Superiority or Other; p = 0.295, Log Rank

5. Secondary Outcome: Propagation Velocity of HAPC
Description: Propagation velocity was calculated as the extension divided by the duration for each HAPC. Mean propagation velocity is the sum of the propagation velocities divided by the number of HAPCs.
Time Frame: over 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm/sec
Arm/Group | Prucalopride | PEG 3350
Number analyzed (Participants) | 9 | 6
cm/sec | 0.467 (0.0803) | 0.646 (0.1074)
Statistical Analysis 1: Comparison: Prucalopride vs PEG 3350; Test type: Superiority or Other; p = 0.180, Linear Mixed-Effect Models Analysis; Mean Difference (Final Values) = -0.179, 95% CI 2-sided [-0.465 to 0.107]

6. Secondary Outcome: Duration of HAPC
Description: The mean duration of all HAPCs was calculated as the sum of the duration of each HAPC divided by the number of HAPCs.
Time Frame: over 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: sec
Arm/Group | Prucalopride | PEG 3350
Number analyzed (Participants) | 9 | 6
sec | 84.9 (8.05) | 69.1 (10.75)
Statistical Analysis 1: Comparison: Prucalopride vs PEG 3350; Test type: Superiority or Other; p = 0.225, Linear Mixed-Effect Models Analysis; Mean Difference (Final Values) = 15.8, 95% CI 2-sided [-12.6 to 44.3]

7. Secondary Outcome: Motility Index
Description: Motility index (mmHg) was summarized for the following 3 time points: pre-dose, 0-5 hours post-dose, and 5-12 hours post-dose. The motility index is defined as the natural logarithm of all peak amplitudes of every contraction +1.
Time Frame: over 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Prucalopride | PEG 3350
Number analyzed (Participants) | 9 | 11
mmHg
  Pre-Dose | 9.467 (0.4668) | 8.312 (0.4403)
  0-5 hours post-dose | 13.661 (0.3221) | 13.349 (0.3520)
  5-12 hours post-dose | 14.208 (0.2976) | 14.390 (0.2489)

ADVERSE EVENTS:
Groups:
- Polyethylene Glycol: 13.8g polyethylene glycol (PEG) 3350 with sodium bicarbonate, sodium chloride, and potassium chloride as a solution in water. Administered twice orally on Day 1 (once in the morning and once prior to lunch).
Arm/Group | Prucalopride | Polyethylene Glycol
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 3/13 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prucalopride (N=13) | Polyethylene Glycol (N=12)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.